CLINICAL TRIAL: NCT04443140
Title: Evaluation of COVID-19 Incidence in Patients With Preeclampsia During Pandemic
Brief Title: Preeclampsia-like Syndrome Induced by COVID-19: Is it a Real Public Health Issue in Pregnancy During the Pandemic?
Status: Completed | Type: Observational
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Resul Karakuş, Medical Doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 70/2020
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Covid-19; Preeclampsia; Pregnancy Related
Keywords: covıd-19; pregnancy; preeclampsia; preeclampsia-like syndrome
MeSH Terms: conditions — COVID-19; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR, lung ultrasound — PCR for Covid-19

SUMMARY:
By applying polymerase chain reaction (PCR) test for Covid-19 to preeclampsia patients who applied to our hospital during the Covid-19 pandemic period, we investigated the frequency of Covid-19 related preeclampsia-like syndrome in this patient group.

DETAILED DESCRIPTION:
The investigators studied the frequency of Covid-19 related preeclampsia-like syndrome by PCR test and lung ultrasound for Covid-19 to preeclampsia patients presenting to the instutution during the Covid-19 pandemic period. The first consecutive 100 preeclampsia patients presented to our hospital during the pandemic will be involved in our study. The primary outcome measure is to detect Covid-19 positivity among the preeclamptic pregnant women..

ELIGIBILITY:
Inclusion Criteria:

* First consecutive 100 pregnant women presenting with preeclamptic symptoms and signs between March 15, 2020 and June 1, 2020.

Exclusion Criteria:

* The pregnancies with known diagnosis of preeclampsia before Covid-19 pandemic
* Preeclamptic patient without a Covid-19 PCR test result
* Pregnant women who does not want to participate in study or does not want their personal informations to be shared
* Pregnant women less than 18 years old and more than 40 years old are excluded

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females are studied.
Study Population: First consecutive 100 preeclamptic pregnant women applied to our hospital during covid-19 pandemic
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
PCR positivity | 3 months
  To detect Covid-19 PCR test positivity among preeclamptic pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Resul Karakus, MD, Principal Investigator — Zeynep Kamil Maternity and Childrens Hospital Training and Research Hospital
Locations (1):
- Zeynep Kamil Maternity and Childrens Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
demographic data of the participants and diagnostic test results will be shared

REFERENCES:
- [Result] Mendoza M, Garcia-Ruiz I, Maiz N, Rodo C, Garcia-Manau P, Serrano B, Lopez-Martinez RM, Balcells J, Fernandez-Hidalgo N, Carreras E, Suy A. Pre-eclampsia-like syndrome induced by severe COVID-19: a prospective observational study. BJOG. 2020 Oct;127(11):1374-1380. doi: 10.1111/1471-0528.16339. Epub 2020 Jun 21. PMID 32479682